CLINICAL TRIAL: NCT02132260
Title: A Multicenter, Double-blind, Randomized, Parallel-group, Placebo-controlled Study to Evaluate the Safety and Efficacy of a Naftifine Hydrochloride Cream 2%and the Naftin® Cream 2% in Patients With Tinea Pedis
Brief Title: Evaluate the Safety and Efficacy of Naftifine Hydrochloride Cream 2% and Naftin® Cream 2% in Patients With Tinea Pedis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFTC 1301
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Tinea Pedis
Keywords: Naftifine; Naftin®; Tinea pedis
MeSH Terms: conditions — Tinea Pedis | interventions — naftifine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Naftifine Hydrochloride Cream 2% (Experimental): Naftifine Hydrochloride Cream 2% (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Naftifine Hydrochloride Cream 2%
- Naftin® Cream 2% (Active Comparator): Naftin® (Naftifine Hydrochloride) Cream 2%
  Interventions: Drug: Naftin® (Naftifine Hydrochloride) Cream 2%
- Placebo Topical Cream (Placebo Comparator): Placebo Topical Cream
  Interventions: Drug: Placebo Topical Cream

INTERVENTIONS:
Drug: Naftifine Hydrochloride Cream 2% — Naftifine Hydrochloride Cream 2% (Taro Pharmaceuticals Inc.) applied once-daily for two weeks
  Other Names: Naftifine
  Arms: Naftifine Hydrochloride Cream 2%
Drug: Naftin® (Naftifine Hydrochloride) Cream 2% — Naftin® (Naftifine Hydrochloride) Cream 2% (Merz Pharmaceuticals, LLC) applied once-daily for two weeks.
  Other Names: Naftifine
  Arms: Naftin® Cream 2%
Drug: Placebo Topical Cream — Placebo Topical Cream (Taro Pharmaceuticals Inc.) applied once-daily for two weeks.
  Other Names: vehicle
  Arms: Placebo Topical Cream

SUMMARY:
The objective of this study is to compare the efficacy and safety of the test formulation of Naftifine Hydrochloride Cream 2% to Naftin® (Naftifine Hydrochloride) 2% Cream in a 6 week study in patients with tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females 18 years or older
* Clinical diagnosis of tinea pedis with lesions localized to the interdigital spaces or predominantly interdigital, but may extend to other areas of the foot
* The presence of interdigital tinea pedis infection
* The sum of the clinical signs and symptoms scores of the target lesion is at least 4, including a minimum score of at least 2 for erythema and a minimum score of 2 for either scaling or pruritus

Exclusion Criteria:

* Females who are pregnant, lactating or planning to become pregnant during the study period
* Use of antipruritics, including antihistamines within 72 hours prior to baseline visit
* Use of topical corticosteroids, antibiotics or antifungal therapies within two weeks prior to baseline visit
* Use of systemic corticosteroids, antibiotics or antifungal therapies within one month prior to baseline visit
* Use of oral terbinafine or itraconazole within two months prior to baseline visit
* Use of immunosuppressive medication or radiation therapy within three months prior to baseline visit
* Any known hypersensitivity to Naftifine Hydrochloride, or any component of the formulation
* Confluent, diffuse moccasin-type tinea pedis of the entire plantar surface
* History of significant or current evidence of chronic infectious disease, system disorder, organ disorder, or other medical condition that would place undue risk by participation or could jeopardize the integrity of study evaluations
* Evidence of any concurrent dermatophytic infection of the toe nails or dermatological condition of the foot that may interfere with tinea pedis evaluation
* Past history of dermatophyte infections with a lack of response ot antifungal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 890 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Therapeutic Cure | 6 weeks
  The proportion of subjects with therapeutic cure (both mycological cure and clinical cure) at the test-of-cure visit conducted four weeks after the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/; Natalie Yantovskiy, Study Director — Taro Pharmaceuticals USA Inc.

IPD SHARING:
Plan to Share IPD: No